CLINICAL TRIAL: NCT01989455
Title: A Single Center, Phase I, Double-blind, Placebo-controlled Evaluation of the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses of Deferiprone Administered by Intravenous Infusion to Healthy Male and Female Volunteers
Brief Title: A Blinded, Placebo-Controlled Study of the Safety and Pharmacokinetics of Single Doses of Intravenous Deferiprone in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ApoPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: LA42-0113
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Healthy Volunteers
Keywords: Healthy; Deferiprone; DFP; L1
MeSH Terms: interventions — Deferiprone; Isoflurophate; Long Interspersed Nucleotide Elements; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (Experimental): Single dose of 500mg deferiprone or placebo administered via intravenous infusion.
  First 2 subjects to enroll: 1 will be randomized to receive deferiprone and the other to receive placebo.
  Next 14 subjects enrolled: 13 will be randomized to receive deferiprone and 1 to receive placebo.
  Interventions: Drug: Deferiprone; Drug: Placebo
- Cohort 2 (Experimental): Single dose of 1000mg deferiprone or placebo administered via intravenous infusion and oral solution.
  Randomization will be done for all 16 subjects at the same time: 14 will be randomized to receive deferiprone and 2 to receive placebo.
  Subjects enrolled to cohort 2 will receive an oral dose of deferiprone.
  Interventions: Drug: Deferiprone; Drug: Placebo
- Cohort 3 (Experimental): Single dose of 1500mg deferiprone or placebo administered via intravenous infusion.
  Randomization will be done for all 16 subjects at the same time, 14 will be randomized to receive deferiprone and 2 to receive placebo.
  Interventions: Drug: Deferiprone; Drug: Placebo
- Cohort 4 (Experimental): Single dose of 2000mg deferiprone or placebo administered via intravenous infusion.
  First 2 subjects to enroll: 1 will be randomized to receive deferiprone and the other to receive placebo.
  Next 14 subjects enrolled: 13 will be randomized to receive deferiprone and 1 to receive placebo.
  Interventions: Drug: Deferiprone; Drug: Placebo

INTERVENTIONS:
Drug: Deferiprone — Deferiprone for infusion, 10mg/mL for intravenous infusion.
  Oral dose of deferiprone: 80mg/mL oral solution. (Cohort 2)
  Other Names: Ferriprox; DFP; L1
Drug: Placebo — Placebo: normal saline solution.
  Other Names: Saline solution.

SUMMARY:
Single center, randomized, double-blind, placebo-controlled, adaptive sequential ascending-dose study for the evaluation of the safety, tolerability, and pharmacokinetics of single doses of deferiprone administered by intravenous infusion to healthy males and females. A bioavailability comparison will be included.

ELIGIBILITY:
Main Inclusion Criteria:

1. Healthy adult males or females, at least 18 years old but not older than 50 years.
2. Body weight at least 60kg.
3. Body Mass Index (BMI) ≥ 18.50 and ≤ 30.00 kg/m2
4. Medically healthy with clinically insignificant screening results (e.g., laboratory profiles, medical history, ECG, vital signs, physical examination.
5. Non or ex-smoker (someone who has completely stopped smoking 6 months before study start)
6. For females, negative result on a serum pregnancy test.

Main Exclusion Criteria:

1. Absolute neutrophil count (ANC) <1.5x10^9/L.
2. History or presence of hypersensitivity to deferiprone or any related products.
3. History or presence of gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs.
4. Presence of significant cardiovascular, pulmonary, hematologic, neurologic, psychiatric, endocrine, immunologic or dermatologic disease.
5. Any history of tuberculosis (TB) or prophylaxis for TB.
6. Suicidal tendency, history of seizures, head trauma with coma or craniotomy/trepanation, state of confusion or relevant psychiatric disease.
7. Inadequate venous access in either arm.
8. Presence of out-of-range cardiac interval or clinically significant ECG abnormalities (PR <110 msec or > 220 msec, QRS <60 msec or >119 msec, QTcB > 450 msec for males and >460 msec for females).
9. Use of acetaminophen, acetylsalicylic acid (ASA), or non-steroidal anti-inflammatory drugs (NSAIDs) in the previous 7 days before study start.
10. Use of any enzyme-modifying drugs, including strong inhibitors of P450 (CYP) enzymes such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem, and HIV antivirals OR strong inducers of CYP enzymes such as: barbiturates, carbamazepine, glucocorticoids, phenytoin, rifampin, and St. John's wart within 28 days prior to study start.
11. Maintenance therapy with any drug, or significant history of drug dependency or alcohol abuse.
12. Had a clinically significant illness during the 28 days prior to study start.
13. Receipt of an investigational product in another clinical trial within 28 days prior prior to study start.
14. Enrolment in a previous cohort of this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Tricta, MD, Study Chair — ApoPharma Inc.
Locations (1):
- Algorithme Pharma Inc., Mount Royal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- 500 mg Deferiprone: Single intravenous dose of 500 mg deferiprone (deferiprone for infusion, 10 mg/mL)
- 1000 mg Deferiprone: Single intravenous dose of 1000 mg deferiprone (deferiprone for infusion, 10 mg/mL), followed one week later by a single oral dose of 1000 mg deferiprone oral solution, 80 mg/mL
- 1500 mg Deferiprone: Single intravenous dose of 1500 mg deferiprone (deferiprone for infusion, 10 mg/mL)
- 2000 mg Deferiprone: Single intravenous dose of 2000 mg deferiprone (deferiprone for infusion, 10 mg/mL)
- Placebo: Single intravenous dose of placebo (normal saline solution).
Period: Overall Study
Arm/Group | 500 mg Deferiprone | 1000 mg Deferiprone | 1500 mg Deferiprone | 2000 mg Deferiprone | Placebo
Started | 14 | 14 | 14 | 14 | 8
Completed | 14 | 12 | 13 | 14 | 7
Not Completed | 0 | 2 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Not completed — Technical problems with infusion | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Healthy volunteers
Groups:
- 500 mg Deferiprone for Infusion: Single intravenous dose of 500 mg deferiprone (deferiprone for infusion, 10 mg/mL)
- 1000 mg Deferiprone for Infusion: Single intravenous dose of 1000 mg deferiprone (deferiprone for infusion, 10 mg/mL)
- 1500 mg Deferiprone for Infusion: Single intravenous dose of 1500 mg deferiprone (deferiprone for infusion, 10 mg/mL)
- 2000 mg Deferiprone for Infusion: Single intravenous dose of 2000 mg deferiprone (deferiprone for infusion, 10 mg/mL)
- Total: Total of all reporting groups
Arm/Group | 500 mg Deferiprone for Infusion | 1000 mg Deferiprone for Infusion | 1500 mg Deferiprone for Infusion | 2000 mg Deferiprone for Infusion | Placebo | Total
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 8 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 14 | 14 | 8 | 64
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 6 | 6 | 4 | 21
  Male | 13 | 10 | 8 | 8 | 4 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 3 | 1 | 8
  White | 12 | 11 | 13 | 11 | 7 | 54
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 14 | 14 | 14 | 14 | 8 | 64

OUTCOME MEASURES:

1. Primary Outcome: Maximum Measured Serum Concentration (Cmax) for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: Cmax was assessed over a 14-hour interval for analyses of deferiprone and its 3-O-glucuronide metabolite in healthy volunteers who received single intravenous doses of 500 mg, 1000 mg, 1500 mg, and 2000 mg of intravenous deferiprone. Blood samples were obtained pre-dose and at 0.17, 0.33, 0.50, 0.75, 1, 1.33, 1.67, 2, 2.5, 3, 4, 6, 9, 12, and 14 hours post-dose.
Time Frame: 14-hour interval
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | 500 mg Deferiprone for Infusion | 1000 mg Deferiprone for Infusion | 1500 mg Deferiprone for Infusion | 2000 mg Deferiprone for Infusion
Number analyzed (Participants) | 14 | 13 | 13 | 14
μg/mL
  Cmax for serum deferiprone | 7.406 (1.889) | 17.835 (2.162) | 27.749 (2.768) | 36.644 (6.643)
  Cmax for serum deferiprone-3-O-glucuronide | 8.037 (1.374) | 16.490 (4.348) | 20.032 (3.757) | 30.517 (3.947)

2. Primary Outcome: Time to Maximum Observed Serum Concentration (Tmax) for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: Tmax was assessed over a 14-hour interval for analyses of deferiprone and its 3-O-glucuronide metabolite in healthy volunteers who received single intravenous doses of 500 mg, 1000 mg, 1500 mg, and 2000 mg of intravenous deferiprone. Blood samples were obtained pre-dose and at 0.17, 0.33, 0.50, 0.75, 1, 1.33, 1.67, 2, 2.5, 3, 4, 6, 9, 12, and 14 hours post-dose.
  The results of the Tmax parameter are reported as the median and range (other parameters are reported as mean and standard deviation).
Time Frame: 14-hour interval
Population: The pharmacokinetic population included all subjects who had sufficient data to derive the value of at least one pharmacokinetic parameter.
Measure: Median (Full Range); unit: hour
Arm/Group | 500 mg Deferiprone for Infusion | 1000 mg Deferiprone for Infusion | 1500 mg Deferiprone for Infusion | 2000 mg Deferiprone for Infusion
Number analyzed (Participants) | 14 | 13 | 13 | 14
hour
  Tmax for Serum Deferiprone | 1.00 [1.00 to 1.33] | 1.00 [0.75 to 1.07] | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Tmax for Serum Deferiprone 3-O-glucuronide | 2.50 [1.67 to 3.00] | 2.50 [1.67 to 3.00] | 2.50 [2.00 to 3.00] | 2.50 [1.67 to 3.00]

3. Primary Outcome: Area Under the Curve From Zero to Infinity (AUC0-∞) for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: AUC0-∞ was assessed over a 14-hour interval for analyses of deferiprone and its 3-O-glucuronide metabolite in healthy volunteers who received single intravenous doses of 500 mg, 1000 mg, 1500 mg, and 2000 mg of intravenous deferiprone. Blood samples were obtained pre-dose and at 0.17, 0.33, 0.50, 0.75, 1, 1.33, 1.67, 2, 2.5, 3, 4, 6, 9, 12, and 14 hours post-dose.
Time Frame: 14-hour interval
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μg*h/mL
Arm/Group | 500 mg Deferiprone for Infusion | 1000 mg Deferiprone for Infusion | 1500 mg Deferiprone for Infusion | 2000 mg Deferiprone for Infusion
Number analyzed (Participants) | 14 | 13 | 14 | 14
μg*h/mL
  AUC0-∞ for serum deferiprone | 18.326 (4.115) | 41.805 (6.797) | 69.390 (8.937) | 89.250 (17.223)
  AUC0-∞ for serum deferiprone 3-O-glucuronide | 38.504 (8.011) | 79.210 (15.686) | 105.829 (13.052) | 161.507 (16.876)

4. Primary Outcome: The Terminal Elimination Half-life (T1/2el) for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: T1/2el was assessed over a 14-hour interval for analyses of deferiprone and its 3-O-glucuronide metabolite in healthy volunteers who received single intravenous doses of 500 mg, 1000 mg, 1500 mg, and 2000 mg of intravenous deferiprone. Blood samples were obtained pre-dose and at 0.17, 0.33, 0.50, 0.75, 1, 1.33, 1.67, 2, 2.5, 3, 4, 6, 9, 12, and 14 hours post-dose.
Time Frame: 14-hour interval
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | 500 mg Deferiprone for Infusion | 1000 mg Deferiprone for Infusion | 1500 mg Deferiprone for Infusion | 2000 mg Deferiprone for Infusion
Number analyzed (Participants) | 14 | 13 | 13 | 14
hour
  T1/2el for serum deferiprone | 1.68 (0.22) | 1.77 (0.32) | 1.83 (0.22) | 1.85 (0.17)
  T1/2el for serum deferiprone 3-O-glucuronide | 2.00 (0.25) | 1.94 (0.25) | 2.01 (0.18) | 1.94 (0.26)

5. Primary Outcome: Safety and Tolerability of Single Ascending Doses of Deferiprone When Administered by Intravenous Infusion in Healthy Volunteers.
Description: The number of participants who experienced adverse events (including any changes of clinical significance in physical examinations, vital signs, 12-lead ECG, and clinical laboratory tests) following a single dose of intravenous deferiprone.
Time Frame: From start of intravenous dosing until Day 5 post-dose for all subjects; and from time of oral dose until 24 hours post-dose for subjects who additionally received oral deferiprone
Population: The safety population included all subjects who received study product.
Measure: Number; unit: participants
Arm/Group | 500 mg Deferiprone for Infusion | 1000 mg Deferiprone for Infusion | 1500 mg Deferiprone for Infusion | 2000 mg Deferiprone for Infusion | Placebo
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 8
participants | 10 | 7 | 8 | 10 | 3

6. Secondary Outcome: Comparison of Cmax for Serum Deferiprone and Deferiprone 3-O-glucuronide Between Deferiprone for Infusion and Oral Deferiprone
Description: Cmax was assessed over a 14-hour interval for deferiprone in healthy volunteers who received a single intravenous dose of 1000 mg and then one week later received a single oral dose of 1000 mg deferiprone oral solution. In both cases, blood samples were obtained pre-dose and at 0.17, 0.33, 0.50, 0.75, 1, 1.33, 1.67, 2, 2.5, 3, 4, 6, 9, 12, and 14 hours post-dose.
Time Frame: 14-hour interval
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μg/mL
Groups:
- 1000 mg Oral Deferiprone: Single oral dose of 1000 mg deferiprone (deferiprone oral solution, 80 mg/mL)
Arm/Group | 1000 mg Deferiprone for Infusion | 1000 mg Oral Deferiprone
Number analyzed (Participants) | 14 | 12
μg/mL
  Cmax for serum deferiprone | 17.835 (2.162) | 11.692 (3.436)
  Cmax for serum deferiprone-3-O-glucuronide | 16.490 (4.348) | 18.806 (5.659)

7. Secondary Outcome: Absolute Bioavailability of Deferiprone
Description: The pharmacokinetic profile was assessed over a 14-hour interval for deferiprone in healthy volunteers who received a single intravenous dose of 1000 mg and then one week later received a single oral dose of 1000 mg deferiprone oral solution. In both cases, blood samples were obtained pre-dose and at 0.17, 0.33, 0.50, 0.75, 1, 1.33, 1.67, 2, 2.5, 3, 4, 6, 9, 12, and 14 hours post-dose.
Time Frame: 14-hour interval
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μg*h/mL
Arm/Group | 1000 mg Deferiprone for Infusion | 1000 mg Oral Deferiprone
Number analyzed (Participants) | 13 | 12
μg*h/mL | 41.805 (6.797) | 30.796 (7.182)
Statistical Analysis 1: Comparison: 1000 mg Deferiprone for Infusion vs 1000 mg Oral Deferiprone; Test type: Superiority or Other; Percent ratio = 73.19, 90% CI 2-sided [68.83 to 77.56]

8. Secondary Outcome: Safety and Tolerability of a Single 1000 mg Oral Dose of Deferiprone
Description: The number of participants who experienced adverse events (including any changes of clinical significance in physical examinations, vital signs, 12-lead ECG, and clinical laboratory tests) following a single dose of oral deferiprone. Note: All subjects in the 1000 mg cohort received active product, including the 2 who had received placebo for the intravenous infusion.
Time Frame: From dosing until 24 hours post-dose
Population: The safety population included all subjects who received study product.
Measure: Number; unit: participants
Arm/Group | 1000 mg Oral Deferiprone
Number analyzed (Participants) | 14
participants | 2

ADVERSE EVENTS:
Arm/Group | 500 mg Deferiprone for Infusion | 1000 mg Deferiprone for Infusion | 1500 mg Deferiprone for Infusion | 2000 mg Deferiprone for Infusion | Placebo | 1000 mg Oral Deferiprone
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14 | 0/8 | 0/14
Other Adverse Events (participants affected / at risk) | 10/14 | 7/14 | 8/14 | 10/14 | 3/8 | 2/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 500 mg Deferiprone for Infusion (N=14) | 1000 mg Deferiprone for Infusion (N=14) | 1500 mg Deferiprone for Infusion (N=14) | 2000 mg Deferiprone for Infusion (N=14) | Placebo (N=8) | 1000 mg Oral Deferiprone (N=14)
Somnolence (Nervous system disorders) | 8 (9) | 5 (5) | 4 (4) | 5 (5) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 4 (4) | 3 (3) | 4 (5) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling of body temperature change (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site swelling (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Generalized erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less